CLINICAL TRIAL: NCT03093688
Title: Phace I and II Study of Immunotherapy Strategy Used iNKT Cells and CD8+T Cells in Patients With Advanced Tumor
Brief Title: Clinical Safty and Efficacy Study of Infusion of iNKT Cells and CD8+T Cells in Patients With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Xiaoyan Zhang, Director of Shanghai Emerging and Re-emerging Infectious Diseases Institute, Shanghai Public Health Clinical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iNKT20170215V1.2
Record Dates: First submitted 2017-03-15; First posted 2017-03-28 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer; Small Cell Lung Cancer; Pancreas Cancer; Hepatocellular Carcinoma; Gastric Cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Pancreatic Neoplasms; Carcinoma, Hepatocellular; Stomach Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: treatment group: receive twice cell infusions in one course of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): The eligible patient receive the experimental infusion of iNKT cells and CD8+T cells .
  Interventions: Biological: Infusion of iNKT cells and CD8+T cells

INTERVENTIONS:
Biological: Infusion of iNKT cells and CD8+T cells — The eligible patients receive twice infusions of iNKT cells(1E8~1E10) and CD8+T cells(1E7~1E9) in one course of treatment.

SUMMARY:
Invariant Natural killer T (iNKT) cells are a unique subset of lymphocytes that express homogeneous TCR recognizing KRN7000 which was up-regulated by many kinds of cancer cells. PD-1+CD8+T cells of patients with advanced tumor are most likely tumor-specified. Our hypothesis is that immunotherapy strategy of infusion of iNKT cells and PD-1+CD8+T cells may decrease the tumor burden and improve overall survival. The purpose of this study is to assess the safety and efficacy of treatment of patients with advanced solid tumor by infusing of iNKT cells and PD-1+CD8+T cells.

DETAILED DESCRIPTION:
Treatment of patients with advance solid tumor is great unsolved challenge to the physicians. Efficacy of conventional treatment, such as surgery, radiotherapy and chemotherapy is limited. AS novel therapy, immunotherapy shows great prospects.

Human iNKT cells can directly lysis tumor cells by a perforin-dependent mechanism,and intracellular granzyme B expression may also potentiate cell killing. Tumor cells expressing CD1d may be especially susceptible to direct NKT cell lysis. iNKT cells play important role in immune regulation by secreting various cytokines. PD-1+CD8+T cells are most likely tumor-specific in patient with advanced tumor. Expansion method of iNKT cells and PD-1+CD8+T cells in vitro is developed as published in our patent. Infusions of iNKT cells and CD8+T cell have been proved safe in mice.

In this clinical trial, the safety and efficacy of the immunotherapy of infusion of iNKT cells and CD8+T cells are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytologically diagnosis of advanced lung cancer, or advanced gastric cancer, or advanced pancrease cancer, or hepatocellular carcinoma, or advanced colorectal cancer
* Patients' tumor tissue (formalin-fixed, paraffin-embedded) must be sufficient for diagnosis of cancer by a certified Laboratory of Pathology
* Laboratory values within the following ranges prior to receiving treatment of study agent: Hemoglobin≧8.0 g/dL, Neutrophils count≧1E9/L, Lymphocytes count≧lower limit of institutional normal, Platelet count≧50E9/L, Serum creatinine≦2.0 mg/dL, Serum bilirubin≦2 x upper limit of institutional normal, AST/ALT≦2 x upper limit of institutional normal
* No dyspnea at rest. Oxygen saturation ≥90% on room air
* No genetic disease
* Fertile females/males must consent to use contraceptives during participation of the trial. Women of child bearing potential must have a negative pregnancy test prior to receiving treatment of study agent within 7 days
* Patients must have a Karnofsky performance status greater than or equal to 80%
* Able and willing to give witnessed, written informed consent form prior to receiving any study related procedure
* Agrees to participate in long-term follow-up for up to 1 years, if received NKT infusion

Exclusion Criteria:

* Organ dysfunction,such as significant cardiovascular disease, myocardial infarction within the past six months, unstable angina, coronary angioplasty within the past six months, uncontrolled atrial or ventricular cardiac arrhythmias; Child-Pugh C; Renal function failure or uremia; Respiratory failure; Disturbance of consciousness; Renal failure.
* Suffering from lymphoma or leukemia
* Serious infections requiring antibiotics, bleeding disorders
* Patients with myelodysplastic syndrome (MDS)
* History of immunodeficiency disease or autoimmune disease
* Positive HIV antigen and antibody, Hepatitis B surface antigen and Hepatitis C PCR within 21 days prior to enrollment
* Within concurrent chemotherapy
* Concurrent other medical condition that would prevent the patient from undergoing protocol-based therapy
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dose of study agent
* Pregnant or breast-feeding patients
* Can't give informed consent
* Lack of availability for follow-up assessment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events related to the infusion of cells | 28 days post-infusion
  The incidence of adverse events following infusion of iNKT cells and CD8+T cells
Objective Response Rate (ORR) | up to 4 months post-infection
  Change of target focus confirmed by CT or MRI

SECONDARY OUTCOMES:
Hematologic analysis | Base line, the day before the first infusion in each course of treatment and up to 12 weeks after the treatment
  Hematologic analysis is used to assess the impact of infusion to the cells in blood, including erythrocytes, leukocytes, platelets, T lymphocytes , B lymphocytes, Natural killer cell, NKT, CD4/CD8, and Treg lymphocytes.
Liver biochemical examination | Base line, the day before the first infusion in each course of treatment and up to 12 weeks after the treatment
  Liver Biochemical examination is a serological analysis about the metabolites related to the function of liver , such as immunoglobulins, Albumin (ALB), Alanine aminotransferase (ALT), Aspartate Aminotransferase (AST), Prealbumin (PA), total bilirubin (TB), and direct bilirubin (DB).
Kidney biochemical examination | Base line, the day before the first infusion in each course of treatment and up to 12 weeks after the treatment
  Kidney Biochemical examination is a serological analysis about the metabolites related to the function of liver, such as Blood urea nitrogen (BUN), Urea (UA), and Crea (Cr).
Tumor Marker | Base line, the day before the first infusion in each course of treatment and up to 12 weeks after the treatment
  Tumor Marker

OTHER OUTCOMES:
Progression-Free Survival (PFS) | Approximately 1 years after the treatment
  Progression-Free Survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Qing J Xu, M.D. Ph.D, Study Chair — Shanghai Public Health Clinical Center
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Cheng X, Jin Y, Xia B, Qin R, Zhang W, Hu H, Mao X, Zhou L, Yan J, Zhang X, Xu J. Safety and Clinical Response to Combined Immunotherapy with Autologous iNKT Cells and PD-1+CD8+ T Cells in Patients Failing First-line Chemotherapy in Stage IV Pancreatic Cancer. Cancer Res Commun. 2023 Jun 7;3(6):991-1003. doi: 10.1158/2767-9764.CRC-23-0137. eCollection 2023 Jun. PMID 37377605
- [Derived] Cheng X, Wang J, Qiu C, Jin Y, Xia B, Qin R, Hu H, Yan J, Zhang X, Xu J. Feasibility of iNKT cell and PD-1+CD8+ T cell-based immunotherapy in patients with lung adenocarcinoma: Preliminary results of a phase I/II clinical trial. Clin Immunol. 2022 May;238:108992. doi: 10.1016/j.clim.2022.108992. Epub 2022 Mar 30. PMID 35367396